CLINICAL TRIAL: NCT00125879
Title: A Long-Term Continuation Study of Patients With Infantile-Onset Pompe Disease Who Were Previously Enrolled in Protocol AGLU01602
Brief Title: Extension Study of Patients With Infantile-Onset Pompe Disease Who Were Previously Enrolled in Protocol AGLU01602
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGLU02403
Record Dates: First submitted 2005-08-01; First posted 2005-08-02 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Glycogen Storage Disease Type II
Keywords: Glycogen Storage Disease Type II; GSD-II; Pompe Disease; Pompe Disease (Late-onset); Acid Maltase Deficiency Disease; Glycogenosis 2; Glycogen Storage Disease Type II (GSD-II)
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Myozyme

INTERVENTIONS:
Biological: Myozyme — 20 mg/kg qow or 40 mg/kg qow
  Other Names: alglucosidase alfa

SUMMARY:
Pompe disease (also known as glycogen storage disease type II) is caused by a deficiency of a critical enzyme in the body called acid alpha-glucosidase (GAA). Normally, GAA is used by the body's cells to break down glycogen (a stored form of sugar) within specialized structures called lysosomes. In patients with Pompe disease, an excessive amount of glycogen accumulates and is stored in various tissues, especially heart and skeletal muscle, which prevents their normal function. The overall objective of this study is to evaluate the long-term safety and efficacy of Myozyme treatment in patients with infantile-onset Pompe disease.

ELIGIBILITY:
Inclusion Criteria:

* The patient's legal guardian(s) must provide written informed consent prior to any study-related procedures being performed
* The patient and his/her legal guardian(s) must have the ability to comply with the clinical protocol
* The patient must have completed Protocol AGLU01602.

Exclusion Criteria:

* Patient has experienced any unmanageable adverse event (AE) in Protocol AGLU01602 due to Myozyme that would preclude continuing treatment with Myozyme

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-06; Primary Completion 2006-06 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Long-term Safety and Efficacy | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (14):
- United States (6):
  - University of Alabama, Birmingham, Alabama
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - Miami Children's Hospital, Miami, Florida
  - Emory University Medical Genetics, Decatur, Georgia
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital Medical Center, Cincinnati, Ohio
- France (2):
  - CHU Amiens, Amiens
  - CHU Cote de Nacre, Caen
- Universitats-Kinderklinik Mainz, Mainz, Germany
- Rambam Medical Center, Haifa, Israel
- San Gerardo Hospital, Monza, Italy
- Erasmus MC University, Rotterdam, Netherlands
- Taiwan (2):
  - Tzu-Chi General Hospital, Hualien City
  - Chi-Mei Medical Center Dept of Pediatrics, Tainan

REFERENCES:
- [Derived] Kishnani PS, Goldenberg PC, DeArmey SL, Heller J, Benjamin D, Young S, Bali D, Smith SA, Li JS, Mandel H, Koeberl D, Rosenberg A, Chen YT. Cross-reactive immunologic material status affects treatment outcomes in Pompe disease infants. Mol Genet Metab. 2010 Jan;99(1):26-33. doi: 10.1016/j.ymgme.2009.08.003. PMID 19775921